CLINICAL TRIAL: NCT04092933
Title: Machine-learning Model for Perioperative Risk Calculation
Brief Title: Perioperative Risk Calculator
Acronym: PROTECT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Technical University of Munich (Other)
Collaborators: Health Information Management, Belgium (Other)
Responsible Party: Sponsor
Other Study IDs: 253/19
Record Dates: First submitted 2019-07-08; First posted 2019-09-17 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-10

CONDITIONS: Perioperative/Postoperative Complications
Keywords: machine learning; decision support; risk calculator; anesthesia
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this project is to develop a machine-learning model for calculating the risk of postoperative complications. In addition to the data collected during the premedication, the model will include all intraoperative values recorded in the Patient Data Management System (PDMS), which include not only vital and respiratory parameters, but also medication and doses, intraoperative events and times. Postoperative complications are defined according to their severity according to the Clavien-Dindo score (Dindo, Demartines et al., 2004) and are collected from the data available in the health information system (HIS).

The machine-learning model is created using an extreme-gradient boosting algorithm which has been updated with new data from the year 2021 to ensure accuracy of the model.

ELIGIBILITY:
Inclusion Criteria:

* all patients who underwent surgery with anesthesia

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent surgical interventions with general or regional anesthesia at Klinikum rechts der Isar, Munich after the implementation of an electronic patient data management system in May 2014
Sampling Method: Non-Probability Sample
Enrollment: 175559 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
postoperative complications | 30 days
  Postoperative complications are classified by means of the Clavien-Dindo-Score.
  The Clavien-Dindo-Score describes classes of severity of postoperative complications:
  Grade I: any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions Grade II: requiring pharmacological treatment Grade IIIa: requiring surgical, endoscopic or radiological intervention not under general anesthesia Grade IIIb: requiring surgical, endoscopic or radiological intervention under general anesthesia Grade IVa: single organ dysfunction Grade IVb: multiorgandysfunction Grade V: death of a patient

SECONDARY OUTCOMES:
in-hospital mortality | 30 days
  mortality within hospital stay

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andonov DI, Ulm B, Graessner M, Podtschaske A, Blobner M, Jungwirth B, Kagerbauer SM. Impact of the Covid-19 pandemic on the performance of machine learning algorithms for predicting perioperative mortality. BMC Med Inform Decis Mak. 2023 Apr 12;23(1):67. doi: 10.1186/s12911-023-02151-1. PMID 37046259